CLINICAL TRIAL: NCT06399991
Title: Aligning Facility Leadership and Climate to Advance Mental Health Services Integration in Malawi (ALIGN)
Brief Title: Aligning Facility Leadership and Climate to Advance Mental Health Services Integration in Malawi
Acronym: ALIGN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-2722; R01MH133028 (NIH)
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted LOCI leadership and climate alignment strategy plus champion strategy (Experimental): Implementation of LOCI strategy (adapted for the Malawian context) plus the champion strategy (enhanced usual care- usual outpatient care enhanced with use of trained champions).
  Interventions: Behavioral: Adapted LOCI leadership and climate alignment strategy plus champion strategy
- Champion strategy (Active Comparator): Enhanced usual care. Continue with usual outpatient care, enhanced with use of trained champions.
  Interventions: Behavioral: Champion strategy

INTERVENTIONS:
Behavioral: Champion strategy — The champion strategy involves identifying champions within each district who are trained and supported as change agents through training and supervision.
  Arms: Champion strategy
Behavioral: Adapted LOCI leadership and climate alignment strategy plus champion strategy — The LOCI strategy involves engaging with district health leadership through data and feedback, leadership development trainings, coaching, and alignment strategy activities to align leadership and climate in support of implementing the evidence-based mental health package. The champion strategy involves identifying champions within each district who are trained and supported as change agents through training and supervision.
  Arms: Adapted LOCI leadership and climate alignment strategy plus champion strategy

SUMMARY:
The main objective of the proposed study is to evaluate the impact of the combined leadership alignment + champion implementation strategy compared to a champion strategy alone, on integration of an evidence-based mental health treatment model into multiple medical care settings.

DETAILED DESCRIPTION:
Task-shared mental health interventions are effective in low- and middle-income countries (LMICs), yet they remain underutilized, and the mental health treatment gap remains substantial. Innovative implementation strategies are needed to successfully integrate evidence-based mental health treatments into medical care in LMICs.

A common component of many implementation efforts is a "champion" strategy which identifies and empowers an on-the-ground staff member as the implementation champion, in charge of focusing their colleagues' efforts on implementation of the evidence-based treatment model. Yet a growing body of research, including our own work in Malawi and elsewhere, highlights that the champion's success is strongly influenced by the strength of support from their line manager and other up-the-chain organization leaders, who are critical in aligning the organization's climate and priorities in support of the implementation effort.

Approaches to influencing leadership engagement to change organizational climate and align priorities has been developed over decades in the field of organizational and industrial psychology but only relatively recently applied to implementation science health research and primarily to implementation in high-income countries. The Leadership and Organizational Change for Implementation (LOCI) is a recently developed multi-level leadership coaching implementation strategy that has demonstrated effectiveness in changing organizational climate, aligning priorities, and enhancing mental health treatment model integration in the US and Norway, but has not been adapted to or tested in low-income country settings. LOCI has significant potential to address the gaps identified in our current research by aligning leadership priorities to support champions in advancing mental health integration.

The overall aim of the proposed study is to evaluate the impact of the combined leadership alignment + champion implementation strategy compared to a champion strategy alone, on integration of an evidence-based mental health treatment model into multiple medical care settings via a cluster-randomized randomized control trial(RCT).

Leadership alignment strategies are an understudied but essential ingredient for successful mental health integration efforts. This project will make a major contribution to our understanding of the role of leadership alignment in advancing evidence-based mental health integration in LMICs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Patient receiving medical care in participating district who screened positive for elevated common mental disorder symptoms that day or in the preceding month.

Exclusion Criteria:

* <18 years old
* Not currently a patient receiving medical care in participating district who screened positive for elevated common mental disorder symptoms that day or in the preceding month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of screening-eligible visits at which patients were screened for mental health | Over the 12 months of the randomized period
  Fidelity of mental health screening will be defined as the proportion of visits eligible for anxiety and depression screening that included the screening. Screening-eligible visits are visits where the patient is not currently receiving mental health treatment. Completion of anxiety and depression screening is defined as completing both the GAD-2 and the Patient Health Questionnaire-2 (PHQ-2), and, if one or both are ≥3, also completing the relevant longer instrument(s) - GAD-7 and PHQ-9. This will be measured utilizing clinical administrative data abstraction.
Proportion of visits at which patients endorsed suicidal ideation at which a suicide risk assessment was completed | Over the 12 months of the randomized period
  Fidelity of safety assessment will be defined as the proportion of patient visits with a PHQ-9 question 9 score >0 that included a documented Suicide Risk Assessment result. This will be measured utilizing clinical administrative data abstraction.
Proportion of patients who were appropriately initiated on mental health treatment | Over the 12 months of the randomized period
  Fidelity of mental health treatment initiation will be defined as the proportion of patients eligible for mental health treatment who actually started either Friendship Bench counseling or medication within 30 days of identification. Eligibility for mental health treatment is defined as having a GAD-7 or PHQ-9 total score of 5 or above. This will be measured utilizing clinical administrative data abstraction.
Proportion of follow-up visits at which clinical decisions followed mental health treatment guidelines | Over the 12 months of the randomized period
  Fidelity of follow-up treatment will be defined as the proportion of follow-up appointments in the first three months of mental health treatment where the clinical treatment decision follows the mental health treatment guidelines. For Friendship Bench (FB) counseling, fidelity is achieved by continuing FB until completion or switching to medication. For medication, if the follow-up GAD-7/PHQ-9 score is <5, fidelity is achieved by continuing treatment; if the follow-up GAD-7/PHQ-9 score is ≥5, fidelity is achieved by continuing treatment and increasing dose. This will be measured utilizing clinical administrative data abstraction.
Proportion of Counseling sessions meeting Fidelity Threshold | Over the 12 months of the randomized period
  Fidelity of Friendship Bench counseling will be defined as the proportion of Friendship Bench counseling sessions receiving a score of ≥3 (Satisfactory) on ≥8 of 10 fidelity checklist items.

SECONDARY OUTCOMES:
Proportion of patients achieving mental health remission | 3 months after participant enrollment
  Mental health remission will be defined as the proportion of patients who achieve depression and anxiety remission at 3 months.
  Anxiety severity is determined using the Generalized Anxiety Disorder scale-7 (GAD-7) which is a seven-item diagnostic tool with total scores ranging from 0 to 21 where higher scores indicate greater self-reported anxiety. Anxiety remission is defined as a score <5.
  Depressive severity is determined using the Patient Health Questionnaire-9 (PHQ-9) which is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression with scores ranging from 0 to 27 where higher scores indicate greater self-reported depression. Depression remission is defined as a score <5.
  Overall remission is defined as both a GAD-7 score <5 and a PHQ-9 score <5, regardless of which score or scores was elevated at baseline.
Proportion of patients achieving chronic condition control | 6 months after participant enrollment
  Chronic condition control will be defined as the proportion of patients whose chronic condition biomarker indicates good control. Patients from the HIV clinic will complete a viral load. Patients from the Non-Communicable Diseases (NCD) clinic will complete a blood pressure measure (hypertension) or HbA1c measure (diabetes). Patients from the Tuberculosis (TB) clinic will complete a sputum smear. Control will be defined for HIV as HIV RNA viral load <1000 c/mL; for hypertension patients as systolic blood pressure <140 mmHg AND diastolic blood pressure <90 mmHg, for diabetes patients as HbA1c < 7.0%; and for TB patients as sputum smear negative.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pence, Principal Investigator — University of North Carolina, Chapel Hill
Locations (12):
- Malawi (12):
  - Chiradzulu District Hospital, Chiradzulu
  - Dedza District Hospital, Dedza
  - Kasungu District Hospital, Kasungu
  - Machinga District Hospital, Machinga
  - Mangochi District Hospital, Mangochi
  - Mchinji District Hospital, Mchinji
  - Mulanje District Hospital, Mulanje
  - Mzimba South District Hospital, Mzimba
  - Nkhata Bay District Hospital, Nkhata Bay
  - Ntcheu District Hospital, Ntcheu
  - Phalombe District Hospital, Phalombe
  - Salima District Hospital, Salima

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data will be uploaded to the National Institute of Mental Health (NIMH) Data Archive (NDA) following a 6-month upload schedule. Data will be available for request from the NDA beginning one year after the grant end date specified on the first Notice of Award. Any subject-level data and the associated analyzed data used in a journal publication will be shared at the time of publication, if the publication occurs before the one-year automatic share date.
Time Frame: All NIMH National Data Archive collection data are shared automatically one year after the grant end date specified on the first Notice of Award.
Access Criteria: Access to data for research purposes will be provided through an NIMH Data Archive Data Access Committee. Investigators and institutions seeking data from NDA will be expected to meet data security measures and will be asked to submit a Data Use Certification, which is cosigned by the investigator and the designated Institutional Official(s) at the NIH-recognized sponsoring institution with a current Federal Wide Assurance.
URL: https://nda.nih.gov/